CLINICAL TRIAL: NCT04171791
Title: A Single Arm, Open-Label Pilot Study of ABT-199 (Venetoclax) for Cutaneous T Cell Lymphoma (CTCL) Stage IB to IV
Brief Title: A Study of ABT-199 (Venetoclax) for Cutaneous T Cell Lymphoma (CTCL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000022803
Record Dates: First submitted 2019-10-29; First posted 2019-11-21 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: CTCL
MeSH Terms: interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ABT-199 (Venetoclax) (Experimental): Patients with Cutaneous T Cell Lymphoma (CTCL) will receive ABT-199 (Venetoclax).
  Interventions: Drug: ABT-199 (venetoclax)

INTERVENTIONS:
Drug: ABT-199 (venetoclax) — Eligible patients will be enrolled into the study and receive venetoclax daily per the US FDA package insert guidelines of venetoclax, with dose escalation up to 400 mg. To minimize the risk of tumor lysis syndrome (TLS), and following the package insert directions for dose escalation over 5 weeks, the initial dose is 20 mg daily, and may be progressively increased as tolerated to 400 mg by week 5.

SUMMARY:
The objective of this study are to evaluate the safety and tolerability of ABT-199 (venetoclax) in patients with advanced Cutaneous T cell lymphoma (CTCL). A secondary objective is to explore clinical response to ABT-199 (venetoclax) in patients with advanced CTCL.

DETAILED DESCRIPTION:
This is a single arm, open-label, non-randomized study with venetoclax (ABT-199) in CTCL patients (subtypes mycosis fungoides and Sézary syndrome only, and excluding transformed mycosis fungoides). This study is planned to be conducted in 18 patients, 18 years or older in age, undergoing a 5-week dose escalation protocol (per the US FDA package insert guidelines of venetoclax for CLL). Safety monitoring will continue throughout the whole period of drug administration and the treatment will be discontinued if intolerable toxicity (defined in Stopping Rules) or disease progression occurs during this period.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed CTCL (subtypes mycosis fungoides and Sézary syndrome only, and excluding transformed mycosis fungoides), stage IB-IV (hereafter referred to as advanced stage). An off-site biopsy report confirming CTCL diagnosis is acceptable.
* All subjects must have shown disease refractory to one or more standard systemic therapy (PUVA, oral bexarotene, vorinostat, romidepsin, and/or Photopheresis) and/or total skin electron beam therapy over 3 months, or have demonstrated relapsed or progressive disease at any time while receiving one or more of therapies.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
* Adequate bone marrow function: WBC > 2000/µL; platelet count > 75,000/mm3; Neutrophil count > 1000/µL, without use of colony stimulating factors (CSF).
* Required washout period for prior therapies

  1. Spot Skin Radiation Therapy (≤10% skin surface): 4 weeks
  2. Systemic therapy: 4 weeks, or until recovered from toxicities
* Women of child-bearing potential must have negative serum pregnancy test and use accepted highly effective methods of birth control throughout the study and for 90 days after dosing and must agree to use effective contraception, such as hormonal birth control (must be at least 3 years without complications), intrauterine devices, double barrier method (condom plus spermicide or diaphragm), or abstain from sexual intercourse.
* Male patients must be willing to use an appropriate method of contraception (e.g., condoms) or abstain from sexual intercourse and inform any sexual partners that they must also use a reliable method of contraception during the study and for 90 days after dosing.
* Adequate hepatic function: bilirubin ≤1.5 x upper limit of normal (ULN), AST ≤3.0 x ULN, ALT ≤ 3.0 x ULN
* Adequate renal function: creatinine clearance ≥ 50 mL/min
* Ability to comply with the treatment schedule

Exclusion Criteria:

* Extracutaneous disease except blood, bone marrow and lymph nodes.
* Concomitant use of any systemic anti-cancer therapy or immune modifier.
* Concomitant use of moderate or strong CYP3A inhibitors or inducers within 1 week of initiation of study drug administration.
* Patients receiving P-gp inhibitors are not eligible for inclusion unless these agents are discontinued for a washout period of 4 weeks. Patients who are taking medications that are narrow window index P-gp substrates (e.g. digoxin, fexofenadine, loperamide, quinidine, talinolol, vinblastine) are not eligible for enrollment.
* Patients with biopsy confirmed transformed MF.
* Prior allogeneic hematopoietic cell transplant.
* Any ongoing infection requiring antibiotics within 2 weeks prior to the start of the study drug, except for antibiotics (e.g. cephalexin) prescribed superficial skin infection.
* Known history of human immunodeficiency virus (HIV), hepatitis B or C.
* History of prior malignancy with the exception of cervical intraepithelial neoplasia, non-melanoma skin cancer, and adequately treated localized prostate carcinoma (PSA <1.0). Patients with a history of other malignancies must have undergone potentially curative therapy and have no evidence of that disease for five years.
* Uncontrolled intercurrent illness, condition, or circumstances that could limit compliance with the study including, but not limited to, the following: acute or chronic graft versus host disease, uncontrolled diabetes mellitus or hypertension, or psychiatric conditions.
* Major surgery within 8 weeks of enrollment.
* Medically significant cardiac event or unstable cardiovascular function defined as:
* Symptomatic ischemia, unstable angina pectoris
* Uncontrolled clinically significant cardiac arrhythmia
* Symptomatic heart failure NYHA Class ≥ 3
* Myocardial infarction or cardiac surgery within 6 months prior to enrollment
* Cerebrovascular event (transient ischemic attack, stroke or CNS bleeding) within the last 12 months.
* Major bleeding within the last 6 months.
* Use of any investigational agents within 30 days prior to enrollment and for the duration of the study.
* Pregnant or lactating.
* Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Body Temperature | Up to 32 weeks
  Safety and tolerability endpoints will be evaluated on the basis of body temperature.
Blood Pressure- Diastolic | Up to 32 weeks
  Safety and tolerability endpoints will be evaluated on the basis of blood pressure.
Blood Pressure- Systolic | Up to 32 weeks
  Safety and tolerability endpoints will be evaluated on the basis of blood pressure.
Pulse Rate | Up to 32 weeks
  Safety and tolerability endpoints will be evaluated on the basis of pulse rate.
Respiratory Rate | Up to 32 weeks
  Safety and tolerability endpoints will be evaluated on the basis of respiratory rate.
Adverse Events | Up to 32 weeks
  Adverse events will be used to measure the study defined outcome:Toxicity. Toxicity (as adverse events) will measured according to the NCI CTCAE (v5.0) for AEs and clinical laboratory profile; AEs will be collected in all patients who received at least one dose of venetoclax and up to four weeks after last dose (Termination visit).

SECONDARY OUTCOMES:
Skin Clinical Response | Up to 32 weeks
  Exploratory skin clinical responses measured by a modified severity-weighted assessment tool (mSWAT).
Duration of Response | Up to 32 weeks
  Duration of response to treatment will be measured in weeks.
Relapse Free and Progression Free Survival | Up to 32 weeks
  Relapse free and progression free survival based on every 4 week follow up after the initial dose until one of the events occurs first: Progressive disease (PD) is documented, another anticancer treatment is administered and/or 28 weeks are completed after the patient's first dose of venetoclax.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Girardi, MD, FAAD, Principal Investigator — Professor of Dermatology Yale University
Locations (1):
- Yale New Haven Hospital / Smilow Cancer Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No